CLINICAL TRIAL: NCT06607445
Title: Evaluation of the Implementation of the Pharmacogenetics and Personalized Medicine Program "MedeA" in the Extremadura Health Service. Population Cohort [MedeA21].
Brief Title: Evaluation of the Implementation of the Pharmacogenetics and Personalized Medicine Program "MedeA" in the Extremadura Health Service.
Acronym: MedeA
Status: Recruiting | Type: Observational
Sponsor: Complejo Hospitalario Universitario de Badajoz (Other)
Responsible Party: Sponsor
Other Study IDs: MedeA21.01
Record Dates: First submitted 2024-09-12; First posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Adverse Drug Event
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (17):
- Lusitania: Primary health care
- Celtici: Oncology
- Vettonia: Mental health
- Turdulia: Internal medicine
- Lácara: Nephrology
- Tartessos: Neurology
- Cancho Roano: Emergencies
- Oretania: Cardiology
- Carpetania: Rheumatology
- Baeturia: Transplants
- Endovélico: Infectious
- Sirona: Clinical pharmacology
- Gaudeamus: University of extremadura
- Sucellus: Urology
- Mnemosyne: Neurology-Vascular
- Paidos: Pediatrics
- Turuñuelo: Pneumology

SUMMARY:
An open longitudinal observational study, non-randomized, which will include the adult population, attended by the SES, in which preference will be given to those patients under treatment with drugs that can produce relevant adverse effects. It is a naturalistic study in which no pharmacological or other type of intervention will be carried out, only the information recommended in the drug data sheet (pharmacogenetic biomarkers, relevant interactions and clinical contraindications) will be provided.

ELIGIBILITY:
Inclusion Criteria:

Patients with a recent diagnosis and who are to be or are being treated according to usual clinical practice, who meet the criteria to participate in the study, read the corresponding information sheet, sign informed consent and agree to participate, provided they meet the following inclusion criteria:

General criteria for all patients:

* Age ≥ 18 years. In case of minors, they may be included, under the following assumptions:
* If the minor is under 12 years of age, participation will require the consent and signature of the informed consent document by both parents (or their guardian).
* If the minor is between 12 and 16 years of age, a proxy informed consent form will be provided and signed by both parents (if both parents are present at the time of the interview) or only one of them (in which case one of the following two conditions must be stated: that the other parent is not present at the time of the interview but does not object to the participation of the minor in the study or that the signatory is the sole legal guardian of the minor).
* Be registered or potentially/have been attended in the Extremadura Health Service.
* Not have language or communication barrier or present disability being totally dependent on another person.

Exclusion Criteria:

* Failure to meet any of the inclusion criteria described above.
* Refusal by the patient to be part of the cohort initially, or to continue to be part of the cohort during follow-up.
* Manifest difficulty for follow-up.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Consecutive sampling is a widely used non-probability sampling that, if performed correctly, can be considered as random sampling. In this case, patients are selected as they come for consultation and as long as they meet the inclusion criteria.
  SES patients are eligible for inclusion in the study, so that a minimum of 3000 participants are expected to be included in the study in order to ensure adequate frequency of genetic polymorphisms of pharmacogenetic relevance. During the Deployment Phase of the Prescription Support Program, it is estimated that an additional 4,000 to 8,000 patients will be included, with a target of 0.1% of the population of Extremadura.
Sampling Method: Non-Probability Sample
Enrollment: 6445 (Estimated)
Dates: Start 2021-05-26 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the implementation of the Pharmacogenetics and Personalized Medicine Program "MedeA" in the Extremadura Health Service. | December 2024
  To analyze the implementation in the clinical routine of a pharmacogenetics and personalized medicine program in SES patients, evaluating the overall impact on the health system, and at the individual level, general modifications in the clinical response and its temporal evolution.

CONTACTS AND LOCATIONS:
Locations (1):
- Complejo Hospitalario Universitario de Badajoz, Badajoz, Spain